CLINICAL TRIAL: NCT02587650
Title: A Phase II Trial of Targeted Kinase Fusion Inhibition in Unresectable Stage III/IV BRAF/NRAS Wild-Type Melanoma
Brief Title: Capmatinib, Ceritinib, Regorafenib, or Entrectinib in Treating Patients With BRAF/NRAS Wild-Type Stage III-IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Adil Daud, Principal Investigator, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14859; NCI-2017-01421 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: ALK Fusion Protein Expression; BRAF wt Allele; Invasive Skin Melanoma; MET Fusion Gene Positive; NRAS wt Allele; NTRK1 Fusion Positive; NTRK2 Fusion Positive; NTRK3 Fusion Positive; RET Fusion Positive; ROS1 Fusion Positive; Stage III Cutaneous Melanoma; Stage IIIA Cutaneous Melanoma; Stage IIIB Cutaneous Melanoma; Stage IIIC Cutaneous Melanoma; Stage IV Cutaneous Melanoma
MeSH Terms: conditions — Noonan Syndrome 6; Melanoma | interventions — capmatinib; ceritinib; entrectinib; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (capmatinib) (Experimental): Patients with MET fusion receive capmatinib PO BID on day 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Capmatinib; Other: Laboratory Biomarker Analysis
- Arm B (ceritinib) (Experimental): Patients with ALK fusion receive ceritinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Ceritinib; Other: Laboratory Biomarker Analysis
- Arm C (regorafenib) (Experimental): Patients with RET or BRAF fusion receive regorafenib PO QD on day 1-21. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Regorafenib
- Arm D (entrectinib) (Experimental): Patients with NTRK1, NTRK2, NTRK3, OR ROS1 fusion receive entrectinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Entrectinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Capmatinib — Given PO
  Other Names: INC-280; INC280; INCB 28060; INCB028060; INCB28060
  Arms: Arm A (capmatinib)
Drug: Ceritinib — Given PO
  Other Names: LDK 378; LDK378; Zykadia
  Arms: Arm B (ceritinib)
Drug: Entrectinib — Given PO
  Other Names: RXDX-101
  Arms: Arm D (entrectinib)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Stivarga
  Arms: Arm C (regorafenib)

SUMMARY:
This phase II trial studies how well capmatinib, ceritinib, regorafenib, or entrectinib work in treating patients with BRAF/NRAS wild-type stage III-IV melanoma. Capmatinib, ceritinib, regorafenib, or entrectinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the clinical activity of tyrosine kinase inhibitors matched to the tumor-specific fusion kinase in patients with metastatic melanoma.

SECONDARY OBJECTIVES:

I. To estimate tumor stability in melanoma patients treated with kinase inhibitors matched to the tumor-specific fusion kinase.

II. To estimate survival in melanoma patients treated with kinase inhibitors matched to the tumor-specific fusion kinase.

III. To examine the safety and tolerability of kinase inhibitors in patients with melanoma with a fusion kinase.

TERTIARY OBJECTIVES:

I. To explore molecular mechanisms of resistance for patients who progress on therapy.

OUTLINE: Patients are assigned to 1 of 4 arms.

ARM A: Patients with MET fusion receive capmatinib orally (PO) twice daily (BID) on day 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.

ARM B: Patients with ALK fusion receive ceritinib PO once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.

ARM C: Patients with RET or BRAF fusion receive regorafenib PO QD on day 1-21. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.

ARM D: Patients with NTRK1, NTRK2, NTRK3, or ROS1 fusion receive entrectinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up within 30 days and then periodically.

ELIGIBILITY:
Inclusion Criteria:

* CAPMATINIB INCLUSION CRITERIA:

  * Ability to understand a written informed consent document, and the willingness to sign it
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-1
  * Life expectancy >= 12 weeks
  * Histologically or cytologically confirmed invasive melanoma
  * Unresectable stage III or stage IV melanoma by clinical or radiographic criteria
  * Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
  * Documentation of absence of activating and targetable BRAF or NRAS point mutations
  * Presence of an oncogenic kinase fusion involving MET, confirmed by assay by a Clinical Laboratory Improvement Act (CLIA)-approved laboratory
  * Prior treatment with at least one Food and Drug Administration (FDA)-approved drug for unresectable/metastatic melanoma; patients who are treatment-naive but who refuse available standard options and prefer to enroll on this study as their first line of treatment after a thorough informed consent process will be eligible at the discretion of the treating physician
  * Resolution of all acute toxic effects (excluding alopecia) of prior radiotherapy, chemotherapy or surgical procedures to Common Terminology Criteria for Adverse Events (CTCAE) v4.03 grade =< 1
  * Absolute neutrophil count >= 1,500/mm^3
  * Platelets >= 75,000/ microliters (mcL)
  * Hemoglobin >= 9 g/dL (transfusions are allowed)
  * Total bilirubin =< 1.5 x upper limit of normal (ULN); patients with Gilbert?s syndrome may be included if total bilirubin =< 3 x ULN or direct bilirubin =< 1.5 x ULN
  * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN if no liver metastases are present? =< 5 x ULN if liver metastases are present
  * Alkaline phosphatase (ALP) =< 5 x ULN
  * Serum amylase =< grade 2 and asymptomatic; patients with grade 1 or 2 serum amylase at the beginning of the study must be confirmed to have no signs and/or symptoms suggesting pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
  * Serum lipase =< ULN
  * Creatinine OR creatinine clearance within normal limits > 40 mL/min (calculated by Cockgraft-Gault) for patients with creatinine levels above ULN
  * Serum potassium, calcium (corrected for serum albumin), magnesium, phosphorus within normal limits with or without supplementation
* CERITINIB INCLUSION CRITERIA:

  * Ability to understand a written informed consent document, and the willingness to sign it
  * ECOG performance status 0-1
  * Life expectancy >= 12 weeks
  * Histologically or cytologically confirmed invasive melanoma
  * Unresectable stage III or stage IV melanoma by clinical or radiographic criteria
  * Measurable disease by RECIST v1.1
  * Documentation of absence of activating and targetable BRAF or NRAS point mutations
  * Presence of an oncogenic kinase fusion involving ALK, confirmed by assay by a CLIA-approved laboratory
  * Prior treatment with at least one FDA-approved drug for unresectable/metastatic melanoma; patients who are treatment-naive but who refuse available standard options and prefer to enroll on this study as their first line of treatment after a thorough informed consent process will be eligible at the discretion of the treating physician
  * Resolution of all acute toxic effects (excluding alopecia) of prior radiotherapy, chemotherapy or surgical procedures to CTCAE v4.03 grade =< 1
  * Absolute neutrophil count >= 1.5 x 10^9/L
  * Platelets >= 75 x 10^9/L
  * Hemoglobin >= 8 g/dL (transfusions are allowed)
  * Total bilirubin =< 1.5 x upper limit of normal (ULN); patients with Gilbert?s syndrome may be included if total bilirubin =< 3 x ULN and direct bilirubin =< 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) =< 3 x ULN if no liver metastases are present? =< 5 x ULN if liver metastases are present
  * Alkaline phosphatase (ALP) =< 5 x ULN
  * Serum amylase =< 2 x ULN
  * Serum lipase =< ULN
  * Fasting plasma glucose =< 175 mg/dL (=< 9.8 mmol/L)
  * Creatinine OR creatinine clearance < 1.5 mg/dL >= 30 mL/min (calculated by Cockgraft-Gault) for patients with creatinine levels above ULN
  * Serum potassium, calcium (corrected for serum albumin), magnesium, phosphorus within normal limits with or without supplementation
* REGORAFENIB INCLUSION CRITERIA:

  * Ability to understand a written informed consent document, and the willingness to sign it
  * ECOG performance status 0-1
  * Life expectancy >= 12 weeks
  * Histologically or cytologically confirmed invasive melanoma
  * Unresectable stage III or stage IV melanoma by clinical or radiographic criteria
  * Measurable disease by RECIST v1.1
  * Documentation of absence of activating and targetable BRAF or NRAS point mutations
  * Presence of an oncogenic kinase fusion involving BRAF or RET, confirmed by assay by a CLIA-approved laboratory
  * Prior treatment with at least one FDA-approved drug for unresectable/metastatic melanoma; patients who are treatment-naive but who refuse available standard options and prefer to enroll on this study as their first line of treatment after a thorough informed consent process will be eligible at the discretion of the treating physician
  * Resolution of all acute toxic effects (excluding alopecia) of prior radiotherapy, chemotherapy or surgical procedures to CTCAE v4.03 grade =< 1
  * Absolute neutrophil count >= 1,500/mm^3
  * Platelets >= 100,000/mm^3
  * Hemoglobin >= 9 g/dL
  * Total bilirubin =< 1.5 x upper limit of normal (ULN); patients with Gilbert?s syndrome may be included if total bilirubin =< 3 x ULN or direct bilirubin =< 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) =< 2.5 x ULN if no liver metastases are present? =< 5 x ULN if liver metastases are present
  * Alkaline phosphatase (ALP) =< 2.5 x ULN if no liver metastases are present; =< 5 x ULN if bone or liver metastases are present
  * Creatinine OR creatinine clearance =< 1.5 x ULN; > 40 mL/min (calculated by Cockgraft-Gault) for patients with creatinine levels above ULN
  * Serum potassium, calcium (corrected for serum albumin), magnesium, phosphorus within normal limits with or without supplementation
  * International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN (patients who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate, provided that no prior evidence of underlying abnormality in coagulation parameters exists; close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is predose as defined by the local standard of care)
* ENTRECTINIB INCLUSION CRITERIA:

  * Ability to understand a written informed consent document, and the willingness to sign it
  * ECOG performance status 0-2
  * Histologically or cytologically confirmed invasive melanoma
  * Unresectable stage III or stage IV melanoma by clinical or radiographic criteria
  * Measurable disease by RECIST v1.1
  * Patients with central nervous system (CNS) involvement, including leptomeningeal carcinomatosis, which is either asymptomatic or previously-treated and controlled, are allowed; the use of seizure prophylaxis is allowed as long as patients are taking non enzyme-inducing anti-epileptic drugs (non-EIAEDs); if patients were previously on EIAEDs and these have been discontinued, they must have been discontinued for at least 2 weeks prior to the start of entrectinib treatment; if patients require an anti-epileptic medication, a CYP3A4 non-EIAED can be used such as levetiracetam, valproic acid, gabapentin, topiramate, or lacosamide; moderate inducers of CYP450, such as dexamethasone or other glucocorticoids, may be used at the discretion of the investigator; patients requiring steroids must be at a stable or decreasing doses for at least 2 weeks prior to the start of entrectinib treatment
  * Documentation of absence of activating and targetable BRAF or NRAS point mutations
  * Presence of an oncogenic kinase fusion involving ROS1 or NTRK1/2/3, confirmed by assay by a CLIA-approved laboratory
  * Prior treatment with at least one FDA-approved drug for unresectable/metastatic melanoma; patients who are treatment-naive but who refuse available standard options and prefer to enroll on this study as their first line of treatment after a thorough informed consent process will be eligible at the discretion of the treating physician
  * Resolution of all acute toxic effects (excluding alopecia) of prior radiotherapy, chemotherapy or surgical procedures to CTCAE v4.03 grade =< 1
  * Absolute neutrophil count >= 1,000/mm^3
  * Platelets >= 75,000/mcL
  * Hemoglobin >= 8 g/dL (transfusions are allowed)
  * Total bilirubin =< 1.5 x upper limit of normal (ULN); patients with Gilbert?s syndrome may be included if total bilirubin =< 3 x ULN or direct bilirubin =< 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) =< 3.0 x ULN if no liver metastases are present? =< 5 x ULN if liver metastases are present
  * Creatinine OR creatinine clearance within normal limits; > 40 mL/min (calculated by Cockgraft-Gault) for patients with creatinine levels above ULN

Exclusion Criteria:

* CAPMATINIB EXCLUSION CRITERIA: Uveal melanoma
* CAPMATINIB EXCLUSION CRITERIA: Current participation in another therapeutic clinical trial
* CAPMATINIB EXCLUSION CRITERIA: Inability to swallow intact tablets or capsules
* CAPMATINIB EXCLUSION CRITERIA: Previously identified allergy or hypersensitivity to components of capmatinib formulation (crospovidone, mannitol, microcrystalline cellulose, povidone, sodium lauryl sulfate, magnesium stearate, colloidal silicon dioxide, and various coating premixes)
* CAPMATINIB EXCLUSION CRITERIA: Diagnosis of concurrent malignancy or previous malignancy within 3 years before study drug administration (exceptions are superficial skin cancers, or any in situ cancers deemed surgically resected, cured and not requiring systemic therapy, and indolent malignancies that currently do not require treatment)
* CAPMATINIB EXCLUSION CRITERIA: Prior treatment with the following antineoplastic therapies within the following time frame:

  * Any prior treatment with capmatinib, crizotinib, or any other cMET or hepatocyte growth factor (HGF) inhibitor
  * Thoracic radiotherapy to lung fields =< 4 weeks prior to starting capmatinib; for all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy =< 2 weeks prior to starting capmatinib; palliative radiotherapy for bone lesions =< 2 weeks prior to starting capmatinib is allowed
  * Receipt of any anticancer or investigational agent within 4 weeks or =< 5 half-lives of the agent (whichever is longer) prior to the first dose of capmatinib; if previous treatment is a monoclonal antibody, then the treatment must be discontinued at least 4 weeks before the first dose of capmatinib
* CAPMATINIB EXCLUSION CRITERIA: Major surgery (e.g., intrathoracic, intraabdominal or intrapelvic) within 4 weeks prior (2 weeks for resection of brain metastases) to starting capmatinib; video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can be enrolled in the study >= 1 week after the procedure
* CAPMATINIB EXCLUSION CRITERIA: Patients receiving treatment with medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of capmatinib treatment and for the duration of the study:

  * Strong and moderate inhibitors of CYP3A4
  * Strong inducers of CYP3A4
  * Proton pump inhibitors (PPI)
* CAPMATINIB EXCLUSION CRITERIA: Patients on unstable or increasing doses of corticosteroids; if patients are on corticosteroids for endocrine deficiencies or tumor-associated symptoms other than CNS related, dose must have been stabilized or decreasing for at least 5 days before first dose of capmatinib
* CAPMATINIB EXCLUSION CRITERIA: Presence or history of carcinomatous meningitis
* CAPMATINIB EXCLUSION CRITERIA: Known symptomatic brain metastases requiring increasing doses of steroid to manage CNS symptoms within 2 weeks prior to study entry

  * Patients with asymptomatic brain metastases may be enrolled at the discretion of the sponsor as long as the patient is stable and has not required increasing dose of steroids to manage CNS symptoms for at least 2 weeks prior to study enrollment
  * Patients requiring seizure prophylaxis must be taking non-enzyme-inducing anti-epileptic drugs (non-EIAED); if patients were previously on EIAEDs and these have been discontinued, they must be discontinued for at least 1 weeks prior to capmatinib administration; if patients re

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Capmatinib): Patients with MET fusion receive capmatinib orally (PO), twice a day (BID) on day 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Capmatinib: Given orally
  Laboratory Biomarker Analysis: Correlative studies
- Arm B (Ceritinib): Patients with ALK fusion receive ceritinib PO once a day (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Ceritinib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm A (Capmatinib) | Arm B (Ceritinib) | Arm C (Regorafenib) | Arm D (Entrectinib)
Started | 0 | 0 | 1 | 0
Completed | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled on this protocol to Arm C (regorafenib). Evaluable patients would be those with baseline staging, treatment for at least 8 weeks, and at least one post-baseline staging scan while on treatment. No participants meet the criteria to be considered evaluable for this protocol.
Groups:
- Arm C (Regorafenib): Participants with RET or BRAF mutations
Arm/Group | Arm C (Regorafenib)
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  60-65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Overall Response Rate (ORR)
Description: Defined as a complete or partial response as per Response Evaluation Criteria in Solid Tumors version 1.1 criteria with confirmatory measurements a minimum of 4 weeks after the response-defining determination. Analysis of study results will include ORR estimations of ALK, NTRK, ROS1, RET, MET, and BRAF rearrangement-positive patients.
Time Frame: 24 weeks
Population: Evaluable participants would be those with baseline staging, treatment for at least 8 weeks, and at least one post-baseline staging scan while on treatment. No participants meet the criteria to be considered evaluable for this analysis.
Groups:
- Arm C (Regorafenib): Patients with RET or BRAF mutations
Arm/Group | Arm C (Regorafenib)
Number analyzed (Participants) | 0

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate is defined as the proportion of patients achieving a complete response (CR) or partial response (PR) or stable disease (SD) for > 24 weeks using the same RECIST 1.1 decision matrix used to calculate ORR. The CBR will be estimated for each arm along with a 95% confidence interval
Time Frame: Up to 2 years
Population: Evaluable patients would be those with baseline staging, treatment for at least 8 weeks, and at least one post-baseline staging scan while on treatment. No participants meet the criteria to be considered evaluable for this analysis.
Arm/Group | Arm C (Regorafenib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall defined as the time from treatment start to the progression or death and overall survival defined as the time from treatment start to death will be estimated using Kaplan-Meier methodology.
Time Frame: From treatment start to death, assessed up to 2 years
Population: as for outcome 2
Arm/Group | Arm C (Regorafenib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) defined as the time from treatment start to the progression or death and overall survival defined as the time from treatment start to death will be estimated using Kaplan-Meier methodology
Time Frame: up to 2 years
Population: as for outcome 2
Arm/Group | Arm C (Regorafenib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Evaluation of the Adverse Effect Profile of Each Kinase Inhibitor
Description: Frequencies of toxicities will be tabulated according to CTCAE v4.03 to assess drug safety and tolerability
Time Frame: Up to 2 years
Population: as for outcome 2
Arm/Group | Arm C (Regorafenib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: Analyses will be performed for all participants having received at least one dose of study drug. Only one participant was enrolled on this trial to Arm C (Regorafenib) for a total of 3 months. Adverse Events reported are for single accrued participant
Arm/Group | Arm C (Regorafenib)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Regorafenib) (N=1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm C (Regorafenib) (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (3)

LIMITATIONS AND CAVEATS:
Only 1 participant was enrolled on this study to Arm C (regorafenib) based on the participants mutation profile. The study was terminated after one accrual due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02587650/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02587650/ICF_001.pdf